CLINICAL TRIAL: NCT06717880
Title: Phase I Study to Evaluate the Safety, Tolerability and Efficacy of IBI363 in Combination With Bevacizumab or Furuitinib in Subjects With Advanced Colorectal Cancer
Brief Title: A Study of IBI363 in Combination With Bevacizumab or Furuitinib in Subjects With Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CIBI363Y101
Record Dates: First submitted 2024-11-11; First posted 2024-12-05 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-12

CONDITIONS: Advanced Malignancies
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): IBI363 Combined with Bevacizumab in Subjects with Advanced Colorectal Cancer
  Interventions: Drug: IBI363 combined with Bevacizumab
- Cohort B (Experimental): IBI363 Combined with Furuitinib in Subjects with Advanced Colorectal Cancer
  Interventions: Drug: IBI363 + Furuitinib

INTERVENTIONS:
Drug: IBI363 combined with Bevacizumab — IBI363 will be administrated on Day 1 of every 2 weeks or every 3 weeks, intravenous injection.
  Bevacizumab, intravenous injection.
  Arms: Cohort A
Drug: IBI363 + Furuitinib — IBI363 Q2W or Q3W IV，Furuitinib po
  Arms: Cohort B

SUMMARY:
A Phase 1 study of IBI363 in combination with Bevacizumab or Furuitinib in Subjects with Advanced Colorectal Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Sign written informed consent and be able to comply with the program's visit schedule and related procedures.
2. Male or female subjects, age 18~75 years.
3. Histologically or cytologically confirmed advanced colorectal cancer.
4. Subjects who have progressed on standard therapy, who are unsuitable for standard therapy, who do not have standard therapy, or who have refused standard therapy.
5. Adequate organ function.
6. At least one measurable lesion (target lesion) per RECIST v1.1.
7. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
8. Life expectancy of 3 months or more.
9. Female subjects of childbearing age or male subjects whose partners are female subjects of childbearing age agree to strictly adopt effective contraceptive measures throughout the entire treatment period and 6 months after the treatment period.

Exclusion Criteria:

1. Women who are pregnant or lactating, or intending to become pregnant before, during, or within 6 months after the last dose of study drug.
2. Active epileptic seizures or active central nervous system (CNS ) metastases and so on.
3. Clinically significant cardiovascular or cerebrovascular disease.
4. Interstitial pneumonia, pulmonary fibrosis, pneumoconiosis, drug-associated pneumonia, and radiation pneumonitis requiring steroid hormone or other therapy, as well as history of severe abnormal lung function or other forms of restrictive lung disease.
5. History of allergies, asthma, atopic dermatitis.
6. Subjects with large amounts of pleural effusion or ascites.
7. Active autoimmune disease requiring systemic therapy within 2 years prior to first dose.
8. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
9. Subjects with known or suspected hypersensitivity to the study drug and any excipients.
10. Subject has a prior history of significant toxicity associated with immune checkpoint inhibitor administration or Bevacizumab that requires permanent discontinuation.
11. Subjects with unresolved > Grade 1 toxicity associated with any prior antineoplastic therapy, with the exception of persistent Grade 2 alopecia, peripheral neuropathy and so on.
12. Active uncontrolled bleeding or known bleeding tendency.
13. Any major surgery within 4 weeks prior to the first dose of study drug.
14. Known positive Human Immunodeficiency Virus (HIV) test, active hepatitis B, hepatitis C (HCV), tuberculosis.
15. Severe/active/uncontrolled infection, infection requiring systemic intravenous antibiotic therapy, or unexplained fever within 2 weeks prior to the first dose of study drug.
16. Diagnosis of another malignancy within 5 years prior to the first dose, exceptions include radically treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or radically resected carcinoma in situ, as well as post-radical localized prostate cancer, and papillary thyroid cancer.
17. Presence of any disease, treatment or laboratory test abnormality, or history or current evidence of substance abuse that, in the judgment of the investigator, may compromise the safety of the subject, interfere with obtaining informed consent, affect subject compliance, or compromise the safety evaluation of the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Event (AE), Treatment-Emergent AE (TEAE), Adverse Event of Special Interest (AESI) and Serious Adverse Event (SAE) | Through out the study (up to 2 years)
  Adverse events will be assessed by investigator(s) according to Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0).

SECONDARY OUTCOMES:
Objective response rate (ORR) | Through out the study (up to 2 years)
  The efficacy of solid tumors was evaluated according to Response Evaluation Criteria in Solid Tumours Version 1.1 (RECIST v1.1).
Time to response (TTR) | Through out the study (up to 2 years)
  The efficacy of solid tumors was evaluated according to RECIST v1.1
disease control rate (DCR) | Through out the study (up to 2 years)
  The efficacy of solid tumors was evaluated according to RECIST v1.1
Duration of response (DoR) | Through out the study (up to 2 years)
  The efficacy of solid tumors was evaluated according to RECIST v1.1
Progression-free survival (PFS) | Through out the study (up to 2 years)
  The efficacy of solid tumors was evaluated according to RECIST v1.1
Overall survival (OS) | Through out the study (up to 2 years)
  The efficacy of solid tumors was evaluated according to RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No